CLINICAL TRIAL: NCT02671630
Title: Computerized Cognitive Training Program for Older Persons With Mild Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yam-Ting Kwok, MD, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NSC 101-2314-B-570-001
Record Dates: First submitted 2016-01-23; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Dementia
Keywords: Cognitive function; Depression; Quality of life; Community-based computerized cognitive training program; Randomized controlled trial
MeSH Terms: conditions — Dementia; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Patients receive only usual hospital care
- Experimental group (Experimental): Patients receive only usual hospital care and community-based computerized cognitive training program
  Interventions: Other: A community-based computerized cognitive training program

INTERVENTIONS:
Other: A community-based computerized cognitive training program — The computer training games included: 1) a phonological loop to train the participants to choose correct song from a list of different songs which can be categorized as people, nature, and musical instrument. The difficulty level progressed from choosing one from two to choosing one from three songs; 2) a visual-spatial sketchpad to train the participants to remember and find the same graphs including vegetable, fruits, daily necessity, and numbers. The difficulty level progressed from finding one pair to three pairs of similar graphs; 3) a central executive system to train the participants to execute dual tasks including conducting dual memory, calculating while listening to music, making phone calls, and matching medication at correct time.
  Arms: Experimental group

SUMMARY:
Little is known about the effects of computerized cognitive training programs on mild dementia patients' health. The purpose of this study was to examine the effects of a community-based computerized cognitive training program.

DETAILED DESCRIPTION:
Little is known about the effects of computerized cognitive training programs on mild dementia patients' health. The purpose of this study was to examine the effects of a community-based computerized cognitive training program.However, most of these studies were not randomized controlled trial and the samples of these studies were mostly healthy older persons, patients with brain injuries, or with moderate and severe dementia. A lack of studies for effects of these programs on patients with mild dementia using randomized controlled trials was found. The purpose of this study was to examine the effects of a community-based computerized cognitive training program.

ELIGIBILITY:
Patients' Inclusion Criteria:

* Aged 65 or older,
* Being diagnosed as having mild dementia by a neurologist, and
* Being able to communicate in Mandarin or Taiwanese.

Patients' Exclusion Criteria:

* Vision or hearing impairment.

Caregivers' (proxy) Inclusion Criteria:

* Living with the dementia patient,
* The family member spending the most time on the patient's care, and
* >20 years old.

Caregivers' (proxy) Exclusion Criteria:

* Terminally ill

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Cognitive Abilities as assessed by Cognitive Abilities Screening Instrument. | 3 months
Memory as assessed by Prospective and Retrospective Memory Questionnaire. | 3 months
Cognitive State as assessed by Mini-Mental State Examination | 3 months

SECONDARY OUTCOMES:
Depression as assessed by Geriatric Depression Scale. | 3 months
Quality of Life as assessed by Chinese Dementia Quality of Life, DQoL. | 3 months